CLINICAL TRIAL: NCT01660607
Title: Phase 1-2 Trial for Patients With Advanced Hematologic Malignancies Undergoing Myeloablative Allogeneic HCT With a T-cell Depleted Graft With Infusion of Conventional T-cells and Regulatory T-cells
Brief Title: Phase 1-2 MAHCT w/ TCell Depleted Graft w/ Simultaneous Infusion Conventional and Regulatory T Cell
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Everett Meyer, Associate Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-21257; SU-09142011-8407 (Other: Stanford University); BMT236 (Other: OnCore); 1R01HL114591-01 (NIH); NCI-2011-03025 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Myeloid Leukemia, Chronic; Acute Myelogenous Leukemia; Myelodysplastic Syndromes (MDS); Lymphoma, Non-Hodgkin; Acute Lymphoblastic Leukemia (ALL); Myeloproliferative Syndrome; Acute Myeloid Leukemia; Acute Leukemia; Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1, Phase I: Low Dose Treg + Tcon (Dose escalation) (Experimental): Participants receive low-dose Treg (1e6 cells/kg) and Tcon (3e6 cells/kg) with CD34+ HSPC.
  Interventions: Biological: CD34+ Hematopoietic Progenitor Cells (HSPC); Biological: Regulatory T-Cells (Treg); Biological: Conventional T-Cells (Tcon)
- Cohort 1A, Phase I: Low Dose Treg + Tcon (Dose escalation) (Experimental): Participants receive low-dose Treg (1e6 cells/kg) and Tcon (1e6 cells/kg) with CD34+ HSPC.
  Interventions: Biological: CD34+ Hematopoietic Progenitor Cells (HSPC); Biological: Regulatory T-Cells (Treg); Biological: Conventional T-Cells (Tcon)
- Cohort 2, Phase 1: Mid Dose Treg + Tcon (Dose escalation) (Experimental): Participants receive low-dose Treg (3e6 cells/kg), Tcon (1e6 cells/kg), and CD34+ HSPC following a conditioning regimen.
  Interventions: Biological: CD34+ Hematopoietic Progenitor Cells (HSPC); Biological: Regulatory T-Cells (Treg); Biological: Conventional T-Cells (Tcon); Procedure: Myeloablative Conditioning Regimen
- Cohort 2A, Phase I: Mid Dose Treg + Tcon (Dose escalation) (Active Comparator): Participants receive low-dose Treg (up to 3e6 cells/kg), Tcon (3e6 cells/kg), and CD34+ HSPC following a conditioning regimen.
  Interventions: Biological: CD34+ Hematopoietic Progenitor Cells (HSPC); Biological: Regulatory T-Cells (Treg); Biological: Conventional T-Cells (Tcon); Procedure: Myeloablative Conditioning Regimen
- Cohort 3, Phase I: High Dose Treg + Tcon (Dose escalation) (Experimental): Participants receive high-dose Treg (3e6 cells/kg), Tcon (3e6 cells/kg), and CD34+ HSPC following a conditioning regimen.
  Interventions: Biological: CD34+ Hematopoietic Progenitor Cells (HSPC); Biological: Regulatory T-Cells (Treg); Biological: Conventional T-Cells (Tcon); Procedure: Myeloablative Conditioning Regimen
- Cohort 3A, Phase I: High Dose Treg + Tcon (Dose escalation) (Experimental): Participants receive high-dose Treg (1e6 cells/kg), Tcon (1e6 cells/kg), and CD34+ HSPC following a conditioning regimen.
  Interventions: Biological: CD34+ Hematopoietic Progenitor Cells (HSPC); Biological: Regulatory T-Cells (Treg); Biological: Conventional T-Cells (Tcon); Procedure: Myeloablative Conditioning Regimen
- Phase 2: Myeloablative HCT Control (Active Comparator): Participants receive standard myeloablative conditioning with CD34+ HSPC and no experimental Treg or Tcon.
  Interventions: Biological: CD34+ Hematopoietic Progenitor Cells (HSPC); Procedure: Myeloablative Conditioning Regimen
- Phase 2 Treg + Tcon with Immunosuppression (Experimental): Participants receive Treg and Tcon therapy with immunosuppressive drugs following myeloablative conditioning.
  Interventions: Biological: CD34+ Hematopoietic Progenitor Cells (HSPC); Biological: Regulatory T-Cells (Treg); Biological: Conventional T-Cells (Tcon); Procedure: Myeloablative Conditioning Regimen
- Phase 2 Treg + Tcon without Immunosuppression (Experimental): Participants receive Treg and Tcon therapy without immunosuppressive drugs following myeloablative conditioning.
  Interventions: Biological: CD34+ Hematopoietic Progenitor Cells (HSPC); Biological: Regulatory T-Cells (Treg); Biological: Conventional T-Cells (Tcon); Procedure: Myeloablative Conditioning Regimen

INTERVENTIONS:
Biological: CD34+ Hematopoietic Progenitor Cells (HSPC) — Purified CD34+ hematopoietic progenitor cells used in transplantation.
Biological: Regulatory T-Cells (Treg) — Highly purified CD4+CD25+CD127-FoxP3+ regulatory T cells to reduce graft-versus-host disease.
  Arms: Cohort 1, Phase I: Low Dose Treg + Tcon (Dose escalation); Cohort 1A, Phase I: Low Dose Treg + Tcon (Dose escalation); Cohort 2, Phase 1: Mid Dose Treg + Tcon (Dose escalation); Cohort 2A, Phase I: Mid Dose Treg + Tcon (Dose escalation); Cohort 3, Phase I: High Dose Treg + Tcon (Dose escalation); Cohort 3A, Phase I: High Dose Treg + Tcon (Dose escalation); Phase 2 Treg + Tcon with Immunosuppression; Phase 2 Treg + Tcon without Immunosuppression
Biological: Conventional T-Cells (Tcon) — Conventional CD3+ T cells used for immune reconstitution and graft enhancement.
  Arms: Cohort 1, Phase I: Low Dose Treg + Tcon (Dose escalation); Cohort 1A, Phase I: Low Dose Treg + Tcon (Dose escalation); Cohort 2, Phase 1: Mid Dose Treg + Tcon (Dose escalation); Cohort 2A, Phase I: Mid Dose Treg + Tcon (Dose escalation); Cohort 3, Phase I: High Dose Treg + Tcon (Dose escalation); Cohort 3A, Phase I: High Dose Treg + Tcon (Dose escalation); Phase 2 Treg + Tcon with Immunosuppression; Phase 2 Treg + Tcon without Immunosuppression
Procedure: Myeloablative Conditioning Regimen — Chemotherapy or total body irradiation used before hematopoietic cell transplantation.
  Arms: Cohort 2, Phase 1: Mid Dose Treg + Tcon (Dose escalation); Cohort 2A, Phase I: Mid Dose Treg + Tcon (Dose escalation); Cohort 3, Phase I: High Dose Treg + Tcon (Dose escalation); Cohort 3A, Phase I: High Dose Treg + Tcon (Dose escalation); Phase 2 Treg + Tcon with Immunosuppression; Phase 2 Treg + Tcon without Immunosuppression; Phase 2: Myeloablative HCT Control

SUMMARY:
This study looks at giving specific types of immune cells, called regulatory T cells and conventional T cells, to patients with blood cancers who are receiving a stem cell transplant. These cells are added back to help the immune system recover and reduce complications after the transplant.

DETAILED DESCRIPTION:
Primary Objectives:

* To determine the efficacy, safety and feasibility of administration of several dose combinations of conventional T cells (Tcon) and regulatory T cells (Treg) in patients undergoing allogeneic hematopoietic cell transplantation (HCT) with HLA matched donors (related or unrelated) using a T cell depleted graft [CD34+ hematopoietic progenitor cells ("CD34+ HSPC")], without immune suppression.
* To determine if concomitant single-agent immunosuppression is needed with fresh Treg cells (phase 2 stage 1) * To determine 1-year GvHD-free relapse-free survival (GRFS) post-HCT (phase 2 stage 2).

Secondary Objectives:

* To determine the 1 year OS in patients undergoing allogeneic HCT with matched donors.
* To measure the incidence and severity of acute and chronic graft vs host disease (GvHD)
* To measure incidence of serious infections

ELIGIBILITY:
Recipient Inclusion Criteria

1. Patients with the following diseases that are histopathologically confirmed are eligible

   * Acute leukemia, primary refractory or beyond CR1, or minimal residual disease (MRD) positivity.
   * High risk acute myeloid leukemia in CR1 with any of the following features:
   * Complex karyotype(≥3 clonal chromosomal abnormalities)
   * Any of the following high risk chromosomal abnormalities:

     * Monosomal karyotype (-5, 5q-, -7, 7q-)
     * t(11q23), t(9;11), inv(3), t(3;3) t(6;9) t(9;22)
     * Normal karyotype with fms-like tyrosine kinase 3 (FLT3)-ITD mutation
   * Other high risk features as determined by molecular studies, or clinical presentation as assessed by the treating physician
   * Chronic myelogenous leukemia (accelerated, blast or second chronic phase)
   * Myelodysplastic syndromes
   * Myeloproliferative syndromes
   * Non-Hodgkin lymphoma with poor risk features not suitable for autologous HCT
2. Age ≥18 yo and ≤ 60 yo for patients in Cohort 1 only. At the start of Cohort 2A and beyond, eligibility will be expanded to allow pediatric patients age ≥ 13 yo.
3. Cardiac ejection fraction ≥ 45%
4. Lung diffusion capacity ≥ 50%
5. Calculated creatinine clearance ≥ 50 cc/min
6. Serum glutamic-pyruvic transaminase( SGPT) and serum glutamic-oxaloacetic transaminase (SGOT) ≤ 3.0 x ULN (Upper limit of normal), unless elevated secondary to disease.
7. Total bilirubin ≤ 2 x ULN (patients with Gilbert's syndrome may be included at the discretion of the PI or where hemolysis has been excluded
8. Availability of a HLA matched donor (related or unrelated) defined by Class I (HLA-A and B) serologic typing (or higher resolution) and Class II (HLA DRB1) molecular typing. An HLA matched donor is defined for this study to be a sibling that is HLA matched 6/6; or an unrelated donor that is HLA matched 6/6 or 5/6. A sibling may be a "half sibling."
9. Karnofsky performance status ≥70%

Recipient Exclusion Criteria

1. Seropositive for any of the following:

   HIV ab; hepatitis B sAg; hepatitis C ab
2. Prior myeloablative therapy or hematopoietic cell transplant
3. Candidate for autologous transplant
4. HIV positive
5. Active uncontrolled bacterial, viral or fungal infection, defined as currently taking antimicrobial therapy and progression of clinical symptoms.
6. Uncontrolled central nervous system (CNS) disease involvement
7. Pregnant or a lactating female
8. Positive serum or urine beta human chorionic gonadotropin (HCG) test in females of childbearing potential within 3 weeks of registration
9. Psychosocial circumstances that preclude the patient being able to go through transplant or participate responsibly in follow up care

Donor Inclusion Criteria

1. Age ≥13 yo and ≤ 75 years
2. Karnofsky performance status of ≥ 70% defined by institutional standards
3. Seronegative for HIV 1 RNA (polymerase chair reaction (PCR); HIV 1 and HIV 2 ab (antibody); HTLV 1 and HTLV 2 ab; PCR+ or sAg (surface antigen) hepatitis B ; or PCR+ or sAg for hepatitis C; negative for the Treponema pallidum antibody Syphilis screen; and negative for HIV 1 and hepatitis C by nucleic acid testing (NAT) within 30 days of apheresis collection. In the case that T pallidum antibody tests are positive, donors must:

   * Be evaluated and show no evidence of syphilis infection of any stage by physical exam and history
   * Have completed effective antibiotic therapy to treat syphilis
   * Have a documented negative non treponemal test (such as RPR) or in the case of a positive non treponemal test must be evaluated by an infectious disease expert to evaluate for alternative causes of test positivity and confirm no evidence of active syphilitic disease
4. Must be 6/6 matched sibling donor as determined by HLA typing
5. Female donors of child-bearing potential must have a negative serum or urine beta-HCG test within three weeks of mobilization
6. Capable of undergoing leukapheresis, have adequate venous access, and be willing to undergo insertion of a central catheter should leukapheresis via peripheral vein be inadequate
7. Agreeable to 2nd donation of Peripheral blood stem cell (PBPC) (or bone marrow harvest) in the event of graft failure
8. The donor or legal guardian greater than 18 years of age, capable of signing an institutional review board (IRB-approved consent form.

Donor Exclusion Criteria

1. Evidence of active infection or viral hepatitis
2. HIV positive
3. Medical, physical, or psychological reason that would place the donor at increased risk for complications from growth factor or leukapheresis
4. Lactating female

Ages: 13 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-02-09 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett Meyer, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine Palo Alto, California, United States, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meyer EH, Pavlova A, Villar-Prados A, Bader C, Xie B, Muffly L, Kim P, Sutherland K, Bharadwaj S, Dahiya S, Frank M, Arai S, Johnston L, Miklos D, Rezvani A, Shiraz P, Sidana S, Shizuru J, Weng WK, Agrawal V, Putnam A, Fernhoff N, Tamarisis J, Lu Y, Pawar RD, McClellan JS, Lowsky R, Negrin RS. Donor regulatory T-cell therapy to prevent graft-versus-host disease. Blood. 2025 May 1;145(18):2012-2024. doi: 10.1182/blood.2024026446. PMID 39792934
- [Derived] Bader CS, Pavlova A, Lowsky R, Muffly LS, Shiraz P, Arai S, Johnston LJ, Rezvani AR, Weng WK, Miklos DB, Frank MJ, Tamaresis JS, Agrawal V, Bharadwaj S, Sidana S, Shizuru JA, Fernhoff NB, Putnam A, Killian S, Xie BJ, Negrin RS, Meyer EH. Single-center randomized trial of T-reg graft alone vs T-reg graft plus tacrolimus for the prevention of acute GVHD. Blood Adv. 2024 Mar 12;8(5):1105-1115. doi: 10.1182/bloodadvances.2023011625. PMID 38091578
- [Derived] Meyer EH, Laport G, Xie BJ, MacDonald K, Heydari K, Sahaf B, Tang SW, Baker J, Armstrong R, Tate K, Tadisco C, Arai S, Johnston L, Lowsky R, Muffly L, Rezvani AR, Shizuru J, Weng WK, Sheehan K, Miklos D, Negrin RS. Transplantation of donor grafts with defined ratio of conventional and regulatory T cells in HLA-matched recipients. JCI Insight. 2019 May 16;4(10):e127244. doi: 10.1172/jci.insight.127244. eCollection 2019 May 16. PMID 31092732

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm/Group Title Cohort 1, Phase I: Low Dose Treg + Tcon (Dose Escalation): Participants receive low-dose Treg (1e6 cells/kg) and Tcon (3e6 cells/kg) with CD34+ HSPC.
  CD34+ Hematopoietic Progenitor Cells (HSPC): Purified CD34+ hematopoietic progenitor cells used in transplantation.
  Regulatory T-Cells (Treg): Highly purified CD4+CD25+CD127-FoxP3+ regulatory T cells to reduce graft-versus-host disease.
  Conventional T-Cells (Tcon): Conventional CD3+ T cells used for immune reconstitution and graft enhancement.
- Phase 2, Stage 1 Treg + Tcon With Immunosuppression (Cohort 2A): Participants receive Treg and Tcon therapy with immunosuppressive drugs following myeloablative conditioning.
  CD34+ Hematopoietic Progenitor Cells (HSPC): Purified CD34+ hematopoietic progenitor cells used in transplantation.
  Regulatory T-Cells (Treg): Highly purified CD4+CD25+CD127-FoxP3+ regulatory T cells to reduce graft-versus-host disease.
  Conventional T-Cells (Tcon): Conventional CD3+ T cells used for immune reconstitution and graft enhancement.
  Myeloablative Conditioning Regimen: Chemotherapy or total body irradiation used before hematopoietic cell transplantation.
- Phase 2, Stage 1 Treg + Tcon Without Immunosuppression (Cohort 2A): Participants receive Treg and Tcon therapy without immunosuppressive drugs following myeloablative conditioning.
  CD34+ Hematopoietic Progenitor Cells (HSPC): Purified CD34+ hematopoietic progenitor cells used in transplantation.
  Regulatory T-Cells (Treg): Highly purified CD4+CD25+CD127-FoxP3+ regulatory T cells to reduce graft-versus-host disease.
  Conventional T-Cells (Tcon): Conventional CD3+ T cells used for immune reconstitution and graft enhancement.
  Myeloablative Conditioning Regimen: Chemotherapy or total body irradiation used before hematopoietic cell transplantation.
- Phase 2, Stage 2 Treg + Tcon With Immunosuppression (Cohort 2A): Participants receive Treg and Tcon therapy with immunosuppressive drugs following myeloablative conditioning.
  CD34+ Hematopoietic Progenitor Cells (HSPC): Purified CD34+ hematopoietic progenitor cells used in transplantation. Regulatory T-Cells (Treg): Highly purified CD4+CD25+CD127-FoxP3+ regulatory T cells to reduce graftversus- host disease. Conventional T-Cells (Tcon): Conventional CD3+ T cells used for immune reconstitution and graft enhancement. Myeloablative Conditioning Regimen: Chemotherapy or total body irradiation used before hematopoietic cell transplantation
Period: Overall Study
Arm/Group | Arm/Group Title Cohort 1, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 1A, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 2, Phase 1: Mid Dose Treg + Tcon (Dose Escalation) | Cohort 2A, Phase I: Mid Dose Treg + Tcon (Dose Escalation) | Cohort 3, Phase I: High Dose Treg + Tcon (Dose Escalation) | Cohort 3A, Phase I: High Dose Treg + Tcon (Dose Escalation) | Phase 2, Stage 1 Treg + Tcon With Immunosuppression (Cohort 2A) | Phase 2, Stage 1 Treg + Tcon Without Immunosuppression (Cohort 2A) | Phase 2, Stage 2 Treg + Tcon With Immunosuppression (Cohort 2A)
Started | 1 | 5 | 0 | 6 | 0 | 0 | 12 | 12 | 32
Day +28 Completed | 1 | 5 | 0 | 6 | 0 | 0 | 12 | 12 | 32
12-Month Follow-Up Completed | 1 | 5 | 0 | 6 | 0 | 0 | 10 | 10 | 26
24-Month Follow-Up Completed | 1 | 5 | 0 | 6 | 0 | 0 | 10 | 10 | 24
Completed | 0 | 2 | 0 | 3 | 0 | 0 | 10 | 10 | 24
Not Completed | 1 | 3 | 0 | 3 | 0 | 0 | 2 | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Phase 2 , Stage 1 Treg + Tcon With Immunosuppression (Cohort 2A): Participants receive Treg and Tcon therapy with immunosuppressive drugs following myeloablative conditioning.
  CD34+ Hematopoietic Progenitor Cells (HSPC): Purified CD34+ hematopoietic progenitor cells used in transplantation.
  Regulatory T-Cells (Treg): Highly purified CD4+CD25+CD127-FoxP3+ regulatory T cells to reduce graft-versus-host disease.
  Conventional T-Cells (Tcon): Conventional CD3+ T cells used for immune reconstitution and graft enhancement.
  Myeloablative Conditioning Regimen: Chemotherapy or total body irradiation used before hematopoietic cell transplantation.
- Phase 2, Phase 2 Treg + Tcon With Immunosuppression (Cohort 2A): Participants receive Treg and Tcon therapy with immunosuppressive drugs following myeloablative conditioning.
  CD34+ Hematopoietic Progenitor Cells (HSPC): Purified CD34+ hematopoietic progenitor cells used in transplantation. Regulatory T-Cells (Treg): Highly purified CD4+CD25+CD127-FoxP3+ regulatory T cells to reduce graftversus- host disease. Conventional T-Cells (Tcon): Conventional CD3+ T cells used for immune reconstitution and graft enhancement. Myeloablative Conditioning Regimen: Chemotherapy or total body irradiation used before hematopoietic cell transplantation
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 1A, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 2A, Phase I: Mid Dose Treg + Tcon (Dose Escalation) | Phase 2 , Stage 1 Treg + Tcon With Immunosuppression (Cohort 2A) | Phase 2, Stage 1 Treg + Tcon Without Immunosuppression (Cohort 2A) | Phase 2, Phase 2 Treg + Tcon With Immunosuppression (Cohort 2A) | Total
Number analyzed (Participants) | 1 | 5 | 6 | 12 | 12 | 32 | 68
Age, Customized [Count of Participants; unit: Participants]
  < 30 | 0 | 1 | 1 | 1 | 2 | 11 | 16
  30 - 39 | 0 | 1 | 1 | 4 | 2 | 2 | 10
  40 - 49 | 1 | 2 | 1 | 2 | 4 | 8 | 18
  50 - 59 | 0 | 1 | 3 | 5 | 3 | 5 | 17
  equal or less than 60 | 0 | 0 | 0 | 0 | 1 | 6 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 6 | 3 | 3 | 16 | 30
  Male | 0 | 4 | 0 | 9 | 9 | 16 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 1 | 3 | 7 | 14
  Not Hispanic or Latino | 1 | 4 | 4 | 11 | 9 | 25 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 1 | 9 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 1 | 4 | 3 | 10 | 8 | 17 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 0 | 2 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 1 | 5 | 6 | 12 | 12 | 32 | 68

OUTCOME MEASURES:

1. Primary Outcome: GvHD Free Relapse Free Survival (GRFS)
Description: GvHD-free is defined as no GvHD symptoms, and relapse free survival is defined as survival at 12 months without relapse.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2, Stage 1: Treg + Tcon With Immunosuppression (Cohort 2A); Phase 2, Stage 2: Treg + Tcon With Immunosuppression (Cohort 2A): Participants receive Treg and Tcon therapy with immunosuppressive drugs following myeloablative conditioning.
- Phase 2, Stage 1: Treg + Tcon Without Immunosuppression (Cohort 2A): Participants receive Treg and Tcon therapy without immunosuppressive drugs following myeloablative conditioning.
Arm/Group | Cohort 1, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 1A, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 2A, Phase I: Mid Dose Treg + Tcon (Dose Escalation) | Phase 2, Stage 1: Treg + Tcon With Immunosuppression (Cohort 2A) | Phase 2, Stage 1: Treg + Tcon Without Immunosuppression (Cohort 2A) | Phase 2, Stage 2: Treg + Tcon With Immunosuppression (Cohort 2A)
Number analyzed (Participants) | 1 | 5 | 6 | 12 | 12 | 32
Participants | 1 | 1 | 0 | 9 | 7 | 26

2. Secondary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT) Within 28 Days
Description: Dose-limiting Toxicity (DLT) was assessed as:
  * Absolute neutrophil count <500/µL, to 28 day
  * Cytokine release syndrome/acute infusion reactions as CTCAE Grade 3 to 5
  * Grade 3 to 4 acute GvHD. GvHD was staged as follows:
    * 1: Skin: rash <25%. Liver: bilirubin (BIL) 2-3mg/dL. Gut: diarrhea (DIA) 500-1000 mL/day
    * 2: Skin: rash 25-50%. Liver: BIL 3-6mg/dL. Gut: DIA 1001-1500 mL/day
    * 3: Skin: rash > 50%. Liver: BIL 6-15mg/dL. Gut: DIA >1501-2000 mL/day
    * 4: Skin: generalized erythroderma. Liver: BIL >15mg/dL. Gut: DIA >2001 mL/day GvHD was graded as follows.
    * 1: Skin Stage 1-2; No Liver stage; No Gut stage
    * 2: Skin Stage 1-3 ; Liver Stage 1; +/- Gut Stage 1
    * 3: Skin Stage 2-3, Liver Stage 2-4; +/- Gut Stage 2-3
    * 4: Skin Stage 2-4; Liver Stage 2-4; +/- Gut Stage 2-4 The outcome is reported as the number of participants who received both Treg and Tcon cell infusions and had DLT events, per treatment level.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2, Phase 2 Treg + Tcon With Immunosuppression (Cohort 2A): Participants receive Treg and Tcon therapy with immunosuppressive drugs following myeloablative conditioning.
Arm/Group | Cohort 1, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 1A, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 2A, Phase I: Mid Dose Treg + Tcon (Dose Escalation) | Phase 2, Stage 1: Treg + Tcon With Immunosuppression (Cohort 2A) | Phase 2, Stage 1: Treg + Tcon Without Immunosuppression (Cohort 2A) | Phase 2, Phase 2 Treg + Tcon With Immunosuppression (Cohort 2A)
Number analyzed (Participants) | 1 | 5 | 6 | 12 | 12 | 32
Participants
  Total DLT Events | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Acute GvHD | 1 | 1 | 0 | 0 | 2 | 1
  Grade 4 Acute GvHD | 0 | 0 | 0 | 0 | 0 | 2
  Grade 3-5 CRS | 0 | 0 | 0 | 0 | 0 | 0
  ANC <500 | 0 | 1 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Overall Survival (OS) at 1 Year
Description: Overall Survival (OS) at 1 year was assessed as the number of participants per treatment level that received the hematopoietic cell transplant (HCT), and remained alive 12 months later.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 1A, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 2A, Phase I: Mid Dose Treg + Tcon (Dose Escalation) | Phase 2, Stage 1: Treg + Tcon With Immunosuppression (Cohort 2A) | Phase 2, Stage 1: Treg + Tcon Without Immunosuppression (Cohort 2A) | Phase 2, Stage 2: Treg + Tcon With Immunosuppression (Cohort 2A)
Number analyzed (Participants) | 1 | 5 | 6 | 12 | 12 | 32
Participants | 0 | 2 | 6 | 11 | 10 | 28

4. Secondary Outcome: Number of Participants With Severity of Chronic Graft-vs-Host Disease (cGvHD) at 24 Months
Description: Incidence and severity of chronic GvHD was assessed in participants who received the hematopoietic cell transplant (HCT) at 24 months.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 1A, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 2A, Phase I: Mid Dose Treg + Tcon (Dose Escalation) | Phase 2, Stage 1: Treg + Tcon With Immunosuppression (Cohort 2A) | Phase 2, Stage 1: Treg + Tcon Without Immunosuppression (Cohort 2A) | Phase 2, Stage 2: Treg + Tcon With Immunosuppression (Cohort 2A)
Number analyzed (Participants) | 1 | 5 | 6 | 12 | 12 | 32
Participants
  Milld cGvHD | 0 | 1 | 1 | 1 | 1 | 6
  Moderate cGvHD | 0 | 1 | 0 | 0 | 3 | 7
  Severe cGvHD | 0 | 0 | 0 | 0 | 1 | 0

5. Secondary Outcome: Number of Participants With Incidence of Serious Infections
Description: The outcome is reported as the number of serious infections per treatment level, in participants who received the hematopoietic cell transplant (HCT).
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 1A, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 2A, Phase I: Mid Dose Treg + Tcon (Dose Escalation) | Phase 2, Stage 1: Treg + Tcon Without Immunosuppression (Cohort 2A) | Phase 2, Stage 2: Treg + Tcon With Immunosuppression (Cohort 2A) | Phase 2, Phase 2 Treg + Tcon With Immunosuppression (Cohort 2A)
Number analyzed (Participants) | 1 | 5 | 6 | 12 | 12 | 32
Participants | 0 | 1 | 6 | 3 | 0 | 2

6. Secondary Outcome: Number of Participants Receiving Concomitant Single-Agent Immunosuppression
Description: During Phase 2, stage 1, concomitant single-agent immunosuppression was assessed as in participants receiving fresh Treg cells.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 1A, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 2A, Phase I: Mid Dose Treg + Tcon (Dose Escalation) | Phase 2, Stage 1: Treg + Tcon With Immunosuppression (Cohort 2A) | Phase 2, Stage 1: Treg + Tcon Without Immunosuppression (Cohort 2A) | Phase 2, Stage 2: Treg + Tcon With Immunosuppression (Cohort 2A)
Number analyzed (Participants) | 1 | 5 | 6 | 12 | 12 | 32
Participants | 0 | 1 | 6 | 12 | 12 | 32

ADVERSE EVENTS:
Time Frame: Up to 2 years
Groups:
- Phase 2, Staage 1 Treg + Tcon With Immunosuppression (Cohort 2A): Participants receive Treg and Tcon therapy with immunosuppressive drugs following myeloablative conditioning.
  CD34+ Hematopoietic Progenitor Cells (HSPC): Purified CD34+ hematopoietic progenitor cells used in transplantation.
  Regulatory T-Cells (Treg): Highly purified CD4+CD25+CD127-FoxP3+ regulatory T cells to reduce graft-versus-host disease.
  Conventional T-Cells (Tcon): Conventional CD3+ T cells used for immune reconstitution and graft enhancement.
  Myeloablative Conditioning Regimen: Chemotherapy or total body irradiation used before hematopoietic cell transplantation.
Arm/Group | Cohort 1, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 1A, Phase I: Low Dose Treg + Tcon (Dose Escalation) | Cohort 2A, Phase I: Mid Dose Treg + Tcon (Dose Escalation) | Phase 2, Staage 1 Treg + Tcon With Immunosuppression (Cohort 2A) | Phase 2, Stage 1 Treg + Tcon Without Immunosuppression (Cohort 2A) | Phase 2, Stage 2 Treg + Tcon With Immunosuppression (Cohort 2A)
All-Cause Mortality (participants affected / at risk) | 1/1 | 3/5 | 2/6 | 3/12 | 2/12 | 6/32
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/5 | 6/6 | 2/12 | 6/12 | 10/32
Other Adverse Events (participants affected / at risk) | 0/1 | 4/5 | 6/6 | 11/12 | 11/12 | 25/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Phase I: Low Dose Treg + Tcon (Dose Escalation) (N=1) | Cohort 1A, Phase I: Low Dose Treg + Tcon (Dose Escalation) (N=5) | Cohort 2A, Phase I: Mid Dose Treg + Tcon (Dose Escalation) (N=6) | Phase 2, Staage 1 Treg + Tcon With Immunosuppression (Cohort 2A) (N=12) | Phase 2, Stage 1 Treg + Tcon Without Immunosuppression (Cohort 2A) (N=12) | Phase 2, Stage 2 Treg + Tcon With Immunosuppression (Cohort 2A) (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CML relapse (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Graft failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute GI and Liver GVHD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Liver GVHD (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epstein-Barr Infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhizomucor/aspergillus/rhizopus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhagic cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Altered mental status (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure secondary to pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin GVHD (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma of the bladder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated INR (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transminitis (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Phase I: Low Dose Treg + Tcon (Dose Escalation) (N=1) | Cohort 1A, Phase I: Low Dose Treg + Tcon (Dose Escalation) (N=5) | Cohort 2A, Phase I: Mid Dose Treg + Tcon (Dose Escalation) (N=6) | Phase 2, Staage 1 Treg + Tcon With Immunosuppression (Cohort 2A) (N=12) | Phase 2, Stage 1 Treg + Tcon Without Immunosuppression (Cohort 2A) (N=12) | Phase 2, Stage 2 Treg + Tcon With Immunosuppression (Cohort 2A) (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (5) | 0 (0) | 7 (8) | 8 (9) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
White blood cell decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital Edema (retinal hemorrhage) (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (8) | 4 (6) | 4 (5) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 5 (6) | 5 (5) | 2 (2) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 3 (3) | 5 (6)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 3 (3)
Vomiting (Emesis) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GI GVHD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rectal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fever (General disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (5) | 4 (5) | 0 (0)
Dysuria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 3 (4)
Fatigue (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blast crisis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Oral candidiasis (Thrush) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcus mitis bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
E coli bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic fistula (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridioides difficile (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
rhinovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
BK virus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HSV1 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coag negative staphylococcus aureus bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epstein-Barr virus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
parainfluenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
fungal pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
invasive fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HHV6 Viremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 2 (3) | 3 (3) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other- Thigh pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 3 (3)
Insomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal pruritis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized edema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DVT (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute skin GVHD (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Aspergillus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus (CMV) infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
syncope (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increase (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythematous rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 4 (6)
hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
platelet count decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT01660607/Prot_SAP_000.pdf